CLINICAL TRIAL: NCT04148508
Title: Assessing and Enhancing Emotional Competence for Well-Being in Young Adults: A Principled, Evidence-based, Mobile-health Approach to Prevent Mental Disorders and Promote Mental Well-being
Brief Title: App-based Mental Health Promotion in Young European Adults
Acronym: ECoWeB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University Ghent (Other); Ludwig-Maximilians - University of Munich (Other); Universitat Jaume I (Other); Audeering GMBH (Industry); Institute of Communications and Computer Systems, Athens, Greece (Other); Monsenso (Industry); University of Oxford (Other); Brno University of Technology (Other); The Fraunhofer-Gesellschaft (Other); University of Geneva, Switzerland (Other); Københavns Universitet (Other); Deutsches Jugendinstitut e.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1819/32
Record Dates: First submitted 2019-09-06; First posted 2019-11-01 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Wellbeing; Mental Disorder
Keywords: Promotion; Prevention; Mobile App; Emotional Competence; Emotional Resiliance; Wellbeing
MeSH Terms: conditions — Mental Disorders | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Phase III superiority parallel 3-arm randomised multi-centre, multinational cohort randomized controlled trials (cmRCT)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Researchers will be blinded to condition. Participants join a cohort and all receive an App, but are not explicitly told which condition they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored Emotional Competence (Experimental): Self-help Tailored Emotional Competence delivered via mobile app
  Interventions: Behavioral: Tailored Emotional Competence Self-help; Behavioral: Self-monitoring
- Cognitive-behavioural Approach (Active Comparator): Self-help cognitive-behavioural approach delivered via mobile app
  Interventions: Behavioral: Cognitive-behavioural Approach; Behavioral: Self-monitoring
- Self-monitoring (Placebo Comparator): Self-help self-monitoring delivered via mobile app
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Tailored Emotional Competence Self-help — The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Arms: Tailored Emotional Competence
Behavioral: Cognitive-behavioural Approach — The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Arms: Cognitive-behavioural Approach
Behavioral: Self-monitoring — Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time

SUMMARY:
The ECoWeB Project aims to develop and disseminate a mobile application (App) to provide engaging and personalized tools and psychological skills to promote emotional wellbeing and prevent mental health problems in adolescents and young adults.

The project team involves 8 European nations (the United Kingdom, Germany, Belgium, Spain, Greece, the Czech Republic, Denmark, and Switzerland) working together in order to improve mental health care and access for adolescents and young adults:

* To use technology as a tool to assess and promote emotional well-being.
* To deliver empirically supported psychological interventions through a smart phone application to address the needs of adolescents and young adults.
* To improve mental well-being and prevent mental health problems in European adolescents and young adults.

The ECoWeb project will consist of 2 RCT's within a longitudinal prospective cohort called ECoWeB-PROMOTE (indicating PROMOTION of well-being and good mental health) and ECoWeB-PREVENT (indicating PREVENTION of general distress, poor mental health and emotional disorders) respectively.

These trials share the same recruitment procedure, interventions, outcomes (including self-report measures of well-being, anxiety, and depression) and design. Both are interested in the promotion of well-being and the prevention of general poor mental health in young people. The key difference is whether the participants are deemed to be at higher or lower risk criteria for poor mental health based on their general emotional competence skills, i.e., for those at low risk, do the interventions further enhance well-being, for those at higher risk, do the interventions prevent the worsening of poor mental health, general stress and distress, as well as enhancing well-being. In all cases the recruitment procedure will be the same, but the inclusion and exclusion criteria are different and the primary outcome measures are different hence they are 2 trials, rather than one, all running within the same cohort.

DETAILED DESCRIPTION:
The effect of the personalised self-help on EC, well-being, risk trajectories, general mental health difficulties, and social, educational, and occupational outcomes, will be evaluated using cohort multiple randomized controlled trials (cmRCTs; Relton et al., 2010). Eligible (healthy) individuals within the prospective cohort meeting relevant criteria will consent to be monitored for a year using a self-help app and web-site assessments. Some of the cohort will be selected at random to be offered additional self-help elements within the app.

It is important to recognise that all participants in the cohort consent at the outset to provide data to be used to assess the benefit of the self-help apps for the outcomes of interest. In a cmRCT, a large observational cohort of participants meeting eligibility criteria is recruited (N) and their outcomes regularly measured. For each RCT, information from the cohort is used to identify all eligible participants (NA). Some eligible participants (nA) are randomly selected and offered the app with self-help components. The outcomes of these randomly selected participants (nA) are then compared with the outcomes of eligible participants not randomly selected; that is, for ECoWeB, those receiving usual practice plus the ECoWeB monitoring through the app (NA-nA).

The cmRCT design has multiple advantages:

(i) it effectively combines a prospective long-term longitudinal cohort with a randomised trial(s): random selection of some participants is equivalent to random allocation of all with respect to generating 2+ groups whose selection and treatment have not been influenced by anyone or anything other than chance and where all known or unknown prognostic factors are distributed evenly at baseline, enabling strong inference about the causal effects of each intervention, whilst retaining key comparison groups that provide information as to the natural history of the condition and to usual care, essential for assessing primary prevention; (ii) consent to "try" a particular intervention is sought only from those offered that intervention, thus replicating the information and consent procedures that exist in routine health care; (iii) because individuals consent in advance to the option of having an intervention offered if eligible, the investigators avoid individuals being knowingly allocated to a "lesser" usual care condition, enhancing recruitment and retention; (iii) there is the facility for multiple RCTs within one cohort; (iv) increased efficiency and representativeness of the sample as longitudinal observational studies typically recruit a greater quantity and more representative sample of participants than RCTs; (v) because the investigators are recruiting from the general population of interested young people and not specifically recruiting individuals with elevated vulnerability or identified problems (and not seeking a clinical population - those with current or past history of psychiatric disorders are excluded), this approach minimises issues of stigmatization by making participation not limited to those with mental health issues but open for all - indeed one goal is that this approach to explore EC will spark interest and dialogue about EC and mental health in young people generally, and communicate how EC is relevant to everyone on a continuum (i.e., an explicitly destigmatizing approach), designed as a public health approach for the general population; (vi) there is no re-use of data and permissions as the cmRCT approach requires that the original consent is for both participation in the cohort and potentially being offered an intervention.

The cmRCT design enables us to:

(i) examine the course of mental well-being and general mental health symptoms over time in higher-risk and lower-risk young people determined on their EC profiles, who are left to their own devices, providing a natural course "baseline" group to assess the trajectory of well-being and symptoms over time and its relationship to EC, and to (ii) test if mobile app based self-help designed to improve EC can change this trajectory. The investigators thus simultaneously test: (a) a central assumption of the EC model that deficits in EC at baseline will predict greater symptoms of poor mental health and reduced mental well-being at 3 and 12 months, controlling for baseline symptoms and well-being; (b) evaluate whether manipulating EC enhances outcomes, enabling strong causal inference.

The ECoWeb project will consist of 2 RCT's called ECoWeB-PROMOTE (indicating PROMOTION of well-being and good mental health) and ECoWeB-PREVENT (indicating PREVENTION of general distress, poor mental health and emotional disorders).

These trials share the same recruitment procedure, interventions, outcomes (including self-report measures of well-being, anxiety, and depression) and design. Both are interested in the promotion of well-being and the prevention of general poor mental health in young people. The key difference is whether the participants are deemed to be at higher or lower risk criteria for poor mental health based on their general emotional competence skills, i.e., for those at low risk, do the interventions further enhance well-being, for those at higher risk, do the interventions prevent the worsening of poor mental health, general stress and distress, as well as enhancing well-being. In all cases the recruitment procedure will be the same, but the inclusion and exclusion criteria are different and the primary outcome measures are different hence they are 2 trials, rather than one, all running within the same cohort.

The ECoWeB-PROMOTE trial will recruit participants not showing elevated risk on their EC profile. The ECoWeB-PROMOTE trial primarily aims to improve and maintain wellbeing in those that are relatively well. A range of indices of poor mental health and wellbeing will be used as outcome measures including wellbeing, depression, anxiety and functioning: Because one index Is needed for the primary outcome, wellbeing on the WEMWBS is the primary outcome measure as potentially most relevant and sensitive for a population that is relatively well.

The ECoWeB-PREVENT trial will recruit participants who have a hypothesized elevated risk of poor mental health based on their EC profile (although they are still well as the investigators are excluding participants with current or past psychiatric disorders) with the primary aim of reducing that risk through the self-help app and promoting well-being (but not selected on clinical diagnoses or symptoms). A range of indices of poor mental health and wellbeing will be used as outcome measures including wellbeing, depression, anxiety and functioning: Because one index Is needed for the primary outcome, depression symptoms (on the Patient health Questionnaire 9) have been selected as the primary outcome, as potentially the most sensitive and important index of poor mental health and distress, and as a strong predictor of future mental illness.

Elevated risk will be determined by an assessment of emotional competence (EC). Participants EC will be assessed by their scores on the emotional competence questionnaires that participants complete at their baseline assessment.

An algorithm is being developed to decide what combination of scores on the EC measures represent high and low risk, based on scoring in the least optimal quartile/tertile against normative data for this age group.

The remit for the Horizon2020 grant scheme is to work towards improving promotion of mental wellbeing and primary prevention of mental disorders, hence the ECoWeB-PREVENT and ECoWeB-PROMOTE trials exclude those with a history of past depression and current depression or a diagnosis of bipolar disorder or psychosis. The sample recruited will therefore be as inclusive as possible across the wider population of 16-22year olds and by definition are not a clinical population.

ELIGIBILITY:
ECoWeB-PROMOTE Trial

Inclusion criteria

1. Aged 16-22, in the UK, Spain, Belgium and Germany.
2. not indicating elevated vulnerability based on the EC profile within the baseline assessment (as described above);
3. basic literacy in English, Spanish, German, or Dutch, as indicated by ability to complete consent and online questionnaires (12year old reading age or better).
4. Ability to provide informed consent
5. Available for the full duration of the study (12 months)
6. Regular access to a relevant smart phone (using android or IOS systems)

Exclusion criteria

1. Meeting criteria on self-report electronic screening questionnaires for any of the following

   1. current episode or past episode of major depressive disorder reported on the LIDAS and PHQ9
   2. any diagnosis of depression
   3. active suicidality; or
   4. any history of severe mental health problem (i.e., bipolar/psychosis);
2. Currently receiving psychological therapy or counselling or antidepressants or other psychiatric medication.
3. Elevated vulnerability on their emotional competence as assessed within the baseline assessment

ECoWeB-PREVENT Trial

Inclusion criteria

1. Aged 16-22, in the UK, Spain, Belgium and Germany
2. screened for elevated vulnerability criteria on their Emotional Competence profile as assessed within the baseline assessment (as described above);
3. basic literacy in English, Spanish, German, or Dutch as indicated by ability to complete consent and online questionnaires (12year old reading age or better).
4. Ability to provide informed consent
5. Available for the full duration of the study (12 months)
6. Regular access to a relevant smart phone (using android or IOS systems)

Exclusion criteria

1. Meeting criteria on self-report electronic screening questionnaires for any of the following

   1. current episode or past episode of major depressive disorder reported on the LIDAS and PHQ9
   2. any diagnosis of depression
   3. active suicidality; or
   4. any history of severe mental health problem (i.e., bipolar/psychosis);
2. Currently receiving psychological therapy or counselling or antidepressants or other psychiatric medication.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3794 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Watkins, PhD, Principal Investigator — University of Exeter
Locations (4):
- Ghent University, Ghent, Belgium
- Ludwig-Maximilians-University (LMU), Munich, Muenchen, Germany
- Universitat Jaume I, Valencia, Castellón, Spain
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant and clinical and economic data reported in publications will be made available through the University of Exeter's Institutional Repository - Open Research Exeter (see https://ore.exeter.ac.uk).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, statistical analysis plan and informed consent form will be uploaded with this registration.
  Data Access: Post-analysis, the final anonymised dataset will preferentially be stored in Open Research Exeter (ORE), the University of Exeter's open access repository. The data will be available from 24 months after trial completion (end of December 2021).
Access Criteria: Access to these data is permitted but controlled through requests made via the repository to a review panel from the trial team, led by the chief investigator, which will assess requests on scientific merit and commercial sensitivity. Although use is permitted, this will be on the basis that the source of the data is acknowledged (including the funder) and it includes reference to the data set 'handle', and a data access agreement is signed, subject to approval by funder.

REFERENCES:
- [Background] Relton C, Torgerson D, O'Cathain A, Nicholl J. Rethinking pragmatic randomised controlled trials: introducing the "cohort multiple randomised controlled trial" design. BMJ. 2010 Mar 19;340:c1066. doi: 10.1136/bmj.c1066. No abstract available. PMID 20304934
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Donnellan MB, Oswald FL, Baird BM, Lucas RE. The mini-IPIP scales: tiny-yet-effective measures of the Big Five factors of personality. Psychol Assess. 2006 Jun;18(2):192-203. doi: 10.1037/1040-3590.18.2.192. PMID 16768595
- [Background] Goldberg, L. R., (1999) A broad-bandwith, public-domain, personality inventory measuring the lower-level facets of several Five-Factor models I. Mervielde, I.J. Deary, F. de Fruyt, F. Ostendorf (Eds.), Personality psychology in Europe, Vol. 7, Tilburg University Press, Tilburg (1999), pp. 7-28
- [Background] Bot M, Middeldorp CM, de Geus EJ, Lau HM, Sinke M, van Nieuwenhuizen B, Smit JH, Boomsma DI, Penninx BW. Validity of LIDAS (LIfetime Depression Assessment Self-report): a self-report online assessment of lifetime major depressive disorder. Psychol Med. 2017 Jan;47(2):279-289. doi: 10.1017/S0033291716002312. Epub 2016 Oct 5. PMID 27702414
- [Background] Carver CS. Generalization, adverse events, and development of depressive symptoms. J Pers. 1998 Aug;66(4):607-19. doi: 10.1111/1467-6494.00026. PMID 9728418
- [Background] Scherer, K.R., Hosoya, G., & Ryser, A. (2019). Modelling the effects of dispositional determinants on the frequency of experiencing depressive mood in the Swiss Household Panel. In preparation.
- [Background] Scherer KR. Evidence for the existence of emotion dispositions and the effects of appraisal bias. Emotion. 2021 Sep;21(6):1224-1238. doi: 10.1037/emo0000861. Epub 2020 Jul 27. PMID 32718175
- [Background] Pekrun, R., Goetz, T., Frenzel, A.C., Barchfield, P., & Perry, R.P. (2011). Measuring emotions in students' learning and performance: The Achievement Emotions Questionnaire (AEQ). Contemp Educ Psychol, 36, 36-48
- [Background] Berenson KR, Gyurak A, Ayduk O, Downey G, Garner MJ, Mogg K, Bradley BP, Pine DS. Rejection sensitivity and disruption of attention by social threat cues. J Res Pers. 2009 Dec 1;43(6):1064-1072. doi: 10.1016/j.jrp.2009.07.007. PMID 20160869
- [Background] Mathews A, Mackintosh B. Induced emotional interpretation bias and anxiety. J Abnorm Psychol. 2000 Nov;109(4):602-15. PMID 11195984
- [Background] Nolen-Hoeksema S, Morrow J. A prospective study of depression and posttraumatic stress symptoms after a natural disaster: the 1989 Loma Prieta Earthquake. J Pers Soc Psychol. 1991 Jul;61(1):115-21. doi: 10.1037//0022-3514.61.1.115. PMID 1890582
- [Background] Hopko DR, Stanley MA, Reas DL, Wetherell JL, Beck JG, Novy DM, Averill PM. Assessing worry in older adults: confirmatory factor analysis of the Penn State Worry Questionnaire and psychometric properties of an abbreviated model. Psychol Assess. 2003 Jun;15(2):173-83. doi: 10.1037/1040-3590.15.2.173. PMID 12847777
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Sekwena, E.K. & Fontaine, J.R.J. (2018). Redefining and assessing emotional understanding based on the componential emotion approach. South African J of Psychol, 48(2), 243-254.
- [Background] Schlegel K, Scherer KR. Introducing a short version of the Geneva Emotion Recognition Test (GERT-S): Psychometric properties and construct validation. Behav Res Methods. 2016 Dec;48(4):1383-1392. doi: 10.3758/s13428-015-0646-4. PMID 26416137
- [Derived] Bear HA, Money C, Watkins E, Fazel M. Incentivising participation in mental health app research: lessons learned from a mixed methods randomised controlled trial. BJPsych Open. 2025 May 19;11(3):e111. doi: 10.1192/bjo.2025.48. PMID 40384016
- [Derived] Bralee E, Mostazir M, Warren FC, Newbold A, Hulme C, Cranston T, Aas B, Bear H, Botella C, Burkhardt F, Ehring T, Fazel M, Fontaine JRJ, Frost M, Garcia-Palacios A, Greimel E, Hossle C, Hovasapian A, Huyghe VEI, Iversen N, Karpouzis K, Lochner J, Molinari G, Pekrun R, Platt B, Rosenkranz T, Scherer KR, Schlegel K, Schuller BW, Schulte-Korne G, Suso-Ribera C, Voigt V, Voss M, Watkins ER. Brief use of behavioral activation features predicts benefits of self-help app on depression symptoms: Secondary analysis of a selective prevention trial in young people. J Consult Clin Psychol. 2025 Apr;93(4):293-306. doi: 10.1037/ccp0000917. PMID 40126557
- [Derived] Watkins ER, Warren FC, Newbold A, Hulme C, Cranston T, Aas B, Bear H, Botella C, Burkhardt F, Ehring T, Fazel M, Fontaine JRJ, Frost M, Garcia-Palacios A, Greimel E, Hossle C, Hovasapian A, Huyghe VEI, Karpouzis K, Lochner J, Molinari G, Pekrun R, Platt B, Rosenkranz T, Scherer KR, Schlegel K, Schuller BW, Schulte-Korne G, Suso-Ribera C, Voigt V, Voss M, Taylor RS. Emotional competence self-help app versus cognitive behavioural self-help app versus self-monitoring app to prevent depression in young adults with elevated risk (ECoWeB PREVENT): an international, multicentre, parallel, open-label, randomised controlled trial. Lancet Digit Health. 2024 Dec;6(12):e894-e903. doi: 10.1016/S2589-7500(24)00148-1. Epub 2024 Oct 4. PMID 39368871
- [Derived] Watkins ER, Warren FC, Newbold A, Hulme C, Cranston T, Aas B, Bear H, Botella C, Burkhardt F, Ehring T, Fazel M, Fontaine JRJ, Frost M, Garcia-Palacios A, Greimel E, Hossle C, Hovasapian A, Huyghe VEI, Karpouzis K, Lochner J, Molinari G, Pekrun R, Platt B, Rosenkranz T, Scherer KR, Schlegel K, Schuller BW, Schulte-Korne G, Suso-Ribera C, Voigt V, Voss M, Taylor RS. Emotional competence self-help mobile phone app versus cognitive behavioural self-help app versus self-monitoring app to promote mental wellbeing in healthy young adults (ECoWeB PROMOTE): an international, multicentre, parallel, open-label, randomised controlled trial. Lancet Digit Health. 2024 Dec;6(12):e904-e913. doi: 10.1016/S2589-7500(24)00149-3. Epub 2024 Oct 4. PMID 39368870
- [Derived] Newbold A, Warren FC, Taylor RS, Hulme C, Burnett S, Aas B, Botella C, Burkhardt F, Ehring T, Fontaine JRJ, Frost M, Garcia-Palacios A, Greimel E, Hoessle C, Hovasapian A, Huyghe V, Lochner J, Molinari G, Pekrun R, Platt B, Rosenkranz T, Scherer KR, Schlegel K, Schulte-Korne G, Suso C, Voigt V, Watkins ER. Promotion of mental health in young adults via mobile phone app: study protocol of the ECoWeB (emotional competence for well-being in Young adults) cohort multiple randomised trials. BMC Psychiatry. 2020 Sep 22;20(1):458. doi: 10.1186/s12888-020-02857-w. PMID 32962684

RESULTS

PARTICIPANT FLOW:
Groups:
- PROMOTE Trial Tailored Emotional Competence: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Plus Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A normal sample not showing symptoms of poor mental wellbeing
- PROMOTE Trial Cognitive-behavioural Approach: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Plus Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A normal sample not showing symptoms of poor mental wellbeing
- PROMOTE Trial Self-monitoring: PROMOTE Trial Self-help: self-monitoring delivered via mobile app
  Only Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A normal sample not showing symptoms of poor mental wellbeing
- PREVENT Trial Tailored Emotional Competence: PREVENT Trial: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Plus Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A sub-clinical sample reporting some symptoms poor mental health
- PREVENT Trial Cognitive Behavioural Approach: PREVENT Trial: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Plus Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A sub-clinical sample reporting some symptoms poor mental health
- PREVENT Trial Self-Monitoring: PREVENT Trial Self-help: self-monitoring delivered via mobile app
  Only Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample: A sub-clinical sample reporting some symptoms poor mental health
Period: Overall Study
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored Emotional Competence | PREVENT Trial Cognitive Behavioural Approach | PREVENT Trial Self-Monitoring
Started | 847 | 841 | 844 | 417 | 423 | 422
1 Month Follow up | 449 | 457 | 475 | 208 | 212 | 209
3 Month Follow up | 425 | 443 | 447 | 178 | 191 | 199
12 Month Follow up | 410 | 426 | 424 | 176 | 174 | 186
Completed | 410 | 426 | 424 | 176 | 174 | 186
Not Completed | 437 | 415 | 420 | 241 | 249 | 236

BASELINE CHARACTERISTICS:
Population: The figures above are the total population for the 2 trials (PROMOTE and PREVENT). Broken down by trial the numbers of participants in each arm was:
  Prevent Trial TEC 417, C-BA 423, S-M 422 Promote Trial TEC 847, C-BA 841, S-M 844
Groups:
- PROMOTE Trial Tailored Emotional Competence: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample did not show symptoms of poor mental health at baseline
- PROMOTE Trial Cognitive-behavioural Approach: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample did not show symptoms of poor mental health at baseline
- PROMOTE Trial Self-monitoring: Self-help self-monitoring delivered via mobile app
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample did not show symptoms of poor mental health at baseline
- PREVENT Trial Tailored: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample did show symptoms of poor mental health at baseline
- PREVENT Trial Cognitive-: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample did show symptoms of poor mental health at baseline
- PREVENT Trial Self-monitoring: Self-help self-monitoring delivered via mobile app
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample did show symptoms of poor mental health at baseline
- Total: Total of all reporting groups
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored | PREVENT Trial Cognitive- | PREVENT Trial Self-monitoring | Total
Number analyzed (Participants) | 847 | 841 | 844 | 417 | 423 | 422 | 3794
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There was a small proportion of participants for whom no exact age data was recorded. These participants did confirm that they were in the 16 to 22 age group in their consent form, however their specific age was not recorded due to a technical fault with our system.
  We have exact age for PROMOTE EC 843, CBT 837, SM 837, PREVENT EC 412, CBT 422, EC 419, however all participants were used in the analysis as all confirmed they were in the 16-22 age group.
  years
    Age: number analyzed (Participants) | 843 | 837 | 837 | 412 | 422 | 419 | 3770
    Age | 19.2 (1.9) | 19.2 (1.9) | 19 (1.8) | 18.8 (2.0) | 18.8 (2.0) | 18.8 (1.9) | 19 (1.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender is recorded as Male, Female, Both or Neither as exclusive categories.
  Participants
    Male | 220 | 191 | 202 | 86 | 74 | 93 | 866
    Female | 621 | 642 | 633 | 323 | 339 | 322 | 2880
    Neither | 3 | 7 | 6 | 4 | 8 | 3 | 31
    Both | 3 | 1 | 3 | 4 | 2 | 4 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — There is a slight difference between the numbers here and the overall total as some participants preferred not to to provide information on their ethnicity. Population: A row including ethnicity unknown has been added for each group so that the figures add up to 100%
  Participants
    White | 752 | 726 | 725 | 349 | 355 | 356 | 3263
    Mixed | 39 | 44 | 52 | 22 | 31 | 26 | 214
    Asian | 23 | 37 | 39 | 23 | 19 | 21 | 162
    Black | 6 | 12 | 7 | 7 | 8 | 7 | 47
    Arab | 9 | 8 | 5 | 5 | 2 | 4 | 33
    Other | 13 | 8 | 11 | 5 | 4 | 4 | 45
    Unknown | 5 | 6 | 5 | 6 | 4 | 4 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 166 | 161 | 155 | 60 | 59 | 59 | 660
  United Kingdom | 254 | 256 | 256 | 138 | 139 | 141 | 1184
  Germany | 288 | 287 | 293 | 77 | 77 | 75 | 1097
  Spain | 139 | 137 | 140 | 142 | 148 | 147 | 853
Baseline Measures for each trial [Mean (Standard Deviation); unit: units on a scale] — Baseline Measure PROMOTE Trial: Warwick-Edinburgh Mental Well Being Scale (WEMWBS). Higher score = better outcomes. Minimum score 0, maximum score 70.
  Baseline Measure PREVENT Trial: Patient Health Questionnaire 9 (PHQ9). Higher Score = worse outcomes. Minimum score 0, maximum score 27. Population: PROMOTE trial 2532 participants has wellness as the primary variable of interest so baseline WEMWBS is reported here.
  PREVENT trial 1262 participants PHQ9 has symptoms of depression as the primary variable of interest, so baseline PHQ9 is reported here.
  These two variable will be the primary outcomes at 3 months, but the figures here are baseline data
  units on a scale
    PROMOTE Trial WEMWBS: number analyzed (Participants) | 847 | 841 | 844 | 0 | 0 | 0 | 2532
    PROMOTE Trial WEMWBS | 52.8 (6.5) | 53.1 (6.6) | 52.6 (6.6) |  |  |  | 52.9 (6.6)
    PREVENT Trial PHQ9: number analyzed (Participants) | 0 | 0 | 0 | 417 | 423 | 422 | 1262
    PREVENT Trial PHQ9 |  |  |  | 7.4 (4.3) | 7.7 (4.3) | 7.6 (4.5) | 7.6 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure PROMOTE Trial: Warwick-Edinburgh Mental Well Being Scale (WEMWBS)
Description: WEMWBS Well-being questionnaire (Tennant et al., 2007; Stewart-Brown et al., 2009) Uni-dimensional scale. Higher scores indicate greater well-being. Scale range 0 to 70 where 70 represents high well-being.
Time Frame: Primary outcome endpoint at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored Emotional Competence | Cognitive-behavioural Approach | Self-monitoring
Number analyzed (Participants) | 425 | 443 | 447
score on a scale | 50.8 (7.9) | 51.3 (7.4) | 50.3 (7.6)

2. Primary Outcome: Primary Outcome Measure PREVENT Trial (PHQ9)
Description: PHQ9 Depression questionnaire (Kroenke et al., 2001). Answered are summed to calculate total score. Scale range 0 to 27 where 27 represents severe depression.
Time Frame: Primary outcome endpoint at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored Emotional Competence | Cognitive-behavioural Approach | Self-monitoring
Number analyzed (Participants) | 178 | 191 | 199
score on a scale | 8.4 (4.8) | 7.7 (4.6) | 8.8 (4.9)

3. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: GAD7 Anxiety questionnaire (Spitzer et al., 2006) Answered are summed to calculate total score. Scale range 0 to 21 where 21 represents high anxiety.
Time Frame: Primary end-point at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PREVENT Trial Tailored Emotional Competence: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time
  Sample did show symptoms of poor mental health at baseline
- PREVENT Trial Cognitive-Behavioural Approach: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample did show symptoms of poor mental health at baseline
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored Emotional Competence | PREVENT Trial Cognitive-Behavioural Approach | PREVENT Trial Self-monitoring
Number analyzed (Participants) | 423 | 442 | 447 | 182 | 192 | 201
score on a scale | 5.4 (4) | 5.3 (3.9) | 5.2 (3.8) | 7.3 (4.5) | 7.1 (4.5) | 7.5 (4.4)

4. Secondary Outcome: Work and Social Adjustment Scale (WSAS)
Description: WSAS Social functioning questionnaire (Mundt et al., 2002). Answered are summed to calculate total score. Scale range 0 to 40 where 40 represents low functionality.
Time Frame: Primary outcome endpoint at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored Emotional Competence | PREVENT Trial Cognitive-Behavioural Approach | PREVENT Trial Self-monitoring
Number analyzed (Participants) | 415 | 432 | 438 | 165 | 184 | 194
score on a scale | 10 (6.6) | 9.3 (6.1) | 9.7 (6.4) | 13.6 (7.1) | 12.2 (7.4) | 14.3 (7.4)

5. Secondary Outcome: Quality of Life (EuroQuol 5D-3L)
Description: Quality of life questionnaire (Herdman et al., 2011). Descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
  EQ-5D-3L:
  Unabbreviated name: EuroQol-5 Dimensions - 3 Levels Construct measured: Health status, health related quality of life Unit of measure: scores on a scale (no units) Score range for overall scale: minimum: -0.594; maximum: 1 Method of calculation: the overall score is calculated using a standard algorithm with established value sets specific to each country Subscales: none Higher scores indicate a better health state.
Time Frame: Primary outcome endpoint at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored Emotional Competence | PREVENT Trial Cognitive-Behavioural Approach | PREVENT Trial Self-monitoring
Number analyzed (Participants) | 414 | 432 | 438 | 165 | 184 | 194
score on a scale | 0.91 (0.17) | 0.91 (0.17) | 0.91 (0.15) | 0.86 (0.19) | 0.89 (0.16) | 0.83 (0.23)

6. Secondary Outcome: Adult Service Use Schedule (ADSUS-adapted)
Description: ADSUS Service Use Questionnaire. 5 with two parts, A) first rating of yes/no presence of service use then B) details around times/nights of service use.
  Version used: ADSUS - Adapted Unabbreviated name: Adult Service Use Schedule - Adapted Construct measured: use of health care services over previous 3 months Unit of measure: total number of health care contacts in previous 3 months Method of calculation: number of contacts with each of a range of 10 different health care contact types (GP contacts; nurse contacts; psychiatrist contacts; mental health therapist contacts; mental health hospital admissions; physical health/other hospital admissions; mental health hospital appointments; physical health/other hospital appointments; A&E attendances; ambulance conveyances) in previous 3 months were recorded; these were summed to produce the total number of contacts across all contact types.
Time Frame: Primary outcome endpoint at 3 months
Population: Population is the number of those completing the 3 month follow up and answering the ADSUS questionnaire. Outcome is the mean number of contacts such as GP/hospital appointments and A and E attendances
Measure: Mean (Standard Deviation); unit: contacts
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored | PREVENT Trial Cognitive- | PREVENT Trial Self-monitoring
Number analyzed (Participants) | 414 | 432 | 438 | 163 | 184 | 194
contacts | 2.5 (8.5) | 2 (4.9) | 2 (3.9) | 3.9 (6.6) | 4.3 (12.5) | 3.7 (10.8)

7. Other Pre Specified Outcome: Adverse Events Questionnaire (AEQ)
Description: AEQ (Carver, 1998) Questionnaire to measure stressful events. 5 point scale with a score of 1-5 for each item. This questionnaire was collected in the research project, but not used in the primary analysis (eg. the PROMOTE and PREVENT trials), so is not reported here.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Lifetime Depression Assessment Self-Report Questionnaire (LIDAS)
Description: LIDAS Depression assessment questionnaire (Bot et al, 2017). Higher scores indicate more depressive symptoms. This measure was used in screening to assess whether participants had previously suffered from an episode of clinical depression.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Process (Mediator)- Impact of Social Appraisal on Emotional Competence
Description: General and Achievement Appraisal: Measures of appraisal will be derived from existing well-validated instruments that use participant ratings in response to multiple scenarios to indirectly assess major appraisal dimensions (e.g., the Emotion-Index; the Coping-Index (Scherer, 2007, p. 109-110) and newly developed instruments (e.g., the Appraisal Bias Questionnaire and the Emotion Disposition Index), shortened into one brief instrument. Associated achievement-related emotions and perceived control will be measured using abbreviated and brief domain-general variants of Achievement Emotions Questionnaire subscales, which have excellent reliability, internal test validity and external test validity (Pekrun et al., 2011, 2017) and of the perceived academic control and perceived academic value scales (Marsh et al., 2016; Pekrun et al., 2007, 2017). Final items will depend on reliability and redundancy between measures in validation studies.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Process (Mediator)- Impact of Rejection Sensitivity on Emotional Competence
Description: Social Appraisal: the Rejection Sensitivity Questionnaire (ARSQ) ARSQ (Berenson et al., 2009) will assess rejection sensitivity as an index of social appraisal needs. 9 scenarios with question A and B, score range 1-6.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Process (Mediator)- Impact of Worry on Emotional Competence
Description: Worry and Rumination: rumination will be assessed using well-validated and established questionnaire measure- the 8-item Penn State Worry Questionnaire-Abbreviated (Kertz et al., 2014). Score range 8 to 40 where higher score is more worry.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Process (Mediator)- Impact of Emotional Recognition on Emotional Competence
Description: Emotional Knowledge and Perception: Adapted, shortened and abbreviated versions of the Geneva Emotion Recognition Test Short, GERT-S 20- Performance-based emotion recognition test (Schlegel, K., & Scherer, K. R., 2016), in which users detect and interpret emotions from the face, voice, and body from 20 short video clips.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Process (Mediator)- Impact of Emotional Understanding on Emotional Competence - Emotional Knowledge and Perception
Description: The Components of Emotion Understanding Test (CEUT-S), CEUT-S (Sekwena & Fontaine, 2017)- Questionnaire measure based on the Componential Emotion Approach) will assess emotional understanding and perception.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Process (Mediator)- Impact of Rumination on Emotional Competence
Description: Rumination will be assessed using well-validated and established questionnaire measure, the 5-item Brooding subscale of the Response Style Questionnaire (RSQ) (Treynor et al., 2003). Score 5-20 where higher score indicates more rummination.
Time Frame: Primary outcome endpoint at 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over a 21 month time period. This was made up of 9 month recruitment window, and a 12 month follow up period.
Description: Participants were followed up by 1, 3 and 12 month online survey where they were asked about any medical treatment including hospitalisations. A serious adverse event was categorised as when a participant reported one of the 2 situations:
  an overnight hospitalisation for a mental health reason and/or transport to hospital by ambulance or an overnight stay caused by self harm/injury or misuse of drugs or alcohol.
Groups:
- PROMOTE Trial Tailored Emotional Competence: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample not reporting symptoms of poor mental health at baseline.
- PROMOTE Trial Cognitive-Behavioural Approach: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample not reporting symptoms of poor mental health at baseline.
- PROMOTE Trial Self-monitoring: Self-help self-monitoring delivered via mobile app
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample not reporting symptoms of poor mental health at baseline.
- PREVENT Trial Tailored Emotional Competence: Self-help Tailored Emotional Competence delivered via mobile app
  Tailored Emotional Competence Self-help: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion. Interventions are personalised to the individual based on emotional competence skills. Intervention is in addition to self-monitoring in the app. Intervention components include selection of 2 from 4 of : targeting worry and rumination; increasing emotional knowledge and perception skills; improving achievement appraisals including attribution retraining and growth mindset; improving social appraisals including positive interpretations of ambiguous social events
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample reporting symptoms of poor mental health at baseline.
- PREVENT Trial Cognitive-Behavioural Approach: Self-help cognitive-behavioural approach delivered via mobile app
  Cognitive-behavioural Approach: The active interventions are all entirely self-help and provide psycho-education, tips, advice and strategies for well-being promotion, based on cognitive-behavioural principles such as increased activity and challenging negative thinking. Interventions are generic and common to all participants. Intervention is in addition to self-monitoring in the app.
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample reporting symptoms of poor mental health at baseline.
- PREVENT Trial Self-monitoring: Self-help self-monitoring delivered via mobile app
  Self-monitoring: Self-monitoring app that involves monitoring emotions and emotional events over time within the app and being able to review emotion over time.
  Sample reporting symptoms of poor mental health at baseline.
Arm/Group | PROMOTE Trial Tailored Emotional Competence | PROMOTE Trial Cognitive-Behavioural Approach | PROMOTE Trial Self-monitoring | PREVENT Trial Tailored Emotional Competence | PREVENT Trial Cognitive-Behavioural Approach | PREVENT Trial Self-monitoring
All-Cause Mortality (participants affected / at risk) | 0/847 | 0/841 | 0/844 | 0/417 | 0/423 | 0/422
Serious Adverse Events (participants affected / at risk) | 5/847 | 8/841 | 1/844 | 8/417 | 15/423 | 8/422
Other Adverse Events (participants affected / at risk) | 37/847 | 46/841 | 66/844 | 42/417 | 56/423 | 49/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMOTE Trial Tailored Emotional Competence (N=847) | PROMOTE Trial Cognitive-Behavioural Approach (N=841) | PROMOTE Trial Self-monitoring (N=844) | PREVENT Trial Tailored Emotional Competence (N=417) | PREVENT Trial Cognitive-Behavioural Approach (N=423) | PREVENT Trial Self-monitoring (N=422)
Hospitalisation for overnight stay (Psychiatric disorders) | 5 (5) | 8 (8) | 1 (1) | 8 (8) | 15 (15) | 8 (8) — Participants hospitalised for mental health reasons for 1 or more nights. None of the participants reported their hospitalisation to be due to the intervention. The hospitalisations were identified by participant self-report at follow up.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMOTE Trial Tailored Emotional Competence (N=847) | PROMOTE Trial Cognitive-Behavioural Approach (N=841) | PROMOTE Trial Self-monitoring (N=844) | PREVENT Trial Tailored Emotional Competence (N=417) | PREVENT Trial Cognitive-Behavioural Approach (N=423) | PREVENT Trial Self-monitoring (N=422)
Participant reported suicide risk at follow up (Psychiatric disorders) | 8 (8) | 4 (4) | 10 (10) | 7 (7) | 10 (10) | 8 (8) — Participant replied yes to questions about either regular thoughts about suicide, intentions to hurt or kill themselves, or plans to harm themselves or end their life (in the previous 2 weeks). This was self-reported at 1m follow up.
Participant reported suicide risk at follow-up (Psychiatric disorders) | 7 (7) | 10 (10) | 19 (19) | 13 (13) | 16 (16) | 17 (17) — Participant replied yes to questions about either regular thoughts about suicide, intentions to hurt or kill themselves, or plans to harm themselves or end their life (in the previous 2 weeks). This was self-reported at 3m follow up.
Participant reported suicide risk at follow-up (Psychiatric disorders) | 22 (22) | 32 (32) | 37 (37) | 22 (22) | 30 (30) | 24 (24) — Participant replied yes to questions about either regular thoughts about suicide, intentions to hurt or kill themselves, or plans to harm themselves or end their life (in the previous 2 weeks). This was self-reported at 12m follow up.

LIMITATIONS AND CAVEATS:
This trial was a cohort randomised cohort trial with two cohorts (Promote: for lower vulnerability participants, primary outcome, WEMWBS; Prevent: for higher vulnerability participants, PHQ9 primary outcome), all other methodology, intervention, measures the same, with each trial to be analysed separately. There was an outage of the treatment app for 1 month because of a fire at server firm, necessitating replenishment of sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04148508/Prot_004.pdf
  • Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT04148508/SAP_005.pdf
  • Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04148508/ICF_006.pdf